CLINICAL TRIAL: NCT06103799
Title: Application of Information-Motivation-Behavioral Model-based Continuity of Care on the Peri-implantitis Recovery in Diabetic Implant Overdenture Patients: A Randomised Controlled Trial
Brief Title: Application of Information-Motivation-Behavioral Model-based Continuity of Care on the Peri-implantitis Recovery in Diabetic Implant Overdenture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Yi Zhou, Principal Investigator, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DHZhejiangU-2023(005)
Record Dates: First submitted 2023-10-19; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Bone Resorption; Diabetes
MeSH Terms: conditions — Bone Resorption; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The information-motivation-behavioral skills (IMB) model, first proposed by Fisher, is composed of three elements-information, motivation, and behavioral skills-and is aimed at transferring patients' behavior into a positive direction, including self-behavior management ability, medication compliance and so on. For diabetic patients with poor adherence, the IMB model of care can be considered.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMB model-based continuity of care (Experimental): Intervention through the IMB model-based continuity of care was focused on three aspects:
  1. Information intervention: (a) instructing patients to follow the official account of the dental implant department and introducing the instructions to use the application, (b) regularly updating the educational content and disseminating detailed knowledge about the prevention and treatment of oral diseases, especially for peri-implantitis.
  2. Motivation intervention: (a) providing an online platform for patients to interact with nurses and doctors, where they can obtain professional answers. (b) assessing the risk factors related to peri-implantitis and diabetes and developing appropriate interventions
  3. Behavioral skills intervention: (a) providing feedback on the correct use of tools and implants and cleaning of the overdentures by observing the cleaning videos that the patients were required to upload.
  Interventions: Behavioral: IMB model-based continuity of care
- routine health education (No Intervention): For the control group, standard care was provided in the form of routine health education regarding various topics, such as proper brushing techniques, use of an oral irrigator, and other auxiliary tools. The patients were followed-up via telephonic interviews to monitor their condition, including usage of the implant and lifestyle changes; the interviews were conducted at 2 weeks, 1 month, 3 months, and 6 months after treatment. Data were collected about oral health, blood glucose control, lifestyle habits, and comorbidities by using the compliance questionnaire. Appropriated health education was provided if there were any concerns such as gingival swelling, plaque accumulation, and elevated blood glucose levels.

INTERVENTIONS:
Behavioral: IMB model-based continuity of care — The information-motivation-behavioral skills (IMB) model, first proposed by Fisher, is composed of three elements-information, motivation, and behavioral skills-and is aimed at transferring patients' behavior into a positive direction, including self-behavior management ability, medication compliance and so on. For diabetic patients with poor adherence, the IMB model of care can be considered.
  Arms: IMB model-based continuity of care

SUMMARY:
The investigators recruited 32 diabetic IOD patients with a total of 110 problematic implants who had completed the treatment for peri-implantitis between January 2021 and March 2023 as research subjects. The patients were randomly assigned to the control group or the experimental group using the random number table. The control group received routine postoperative medical advice, whereas the experimental group was given an IMB model-based continuity of care.

DETAILED DESCRIPTION:
Continuity of care involves a series of actions designed to ensure that patients undergoing a transfer from different health care settings (e.g., from hospital to home) or within the same setting (e.g., different units in the hospital) receive different levels of collaborative and continuous care, including discharge planning, referrals, and continuous follow-up and guidance after the patient returns home . It encompasses the roles of both provider and receiver. Patients who actively participate will receive more substantial treatment. Additionally, a retrospective cohort study has shown that continuity of care is associated with lower risk of cardiovascular disease risk among individuals with type 2 diabetes. Another prospective cohort has shown that the application of continuity of care in the dental field enhances oral anticancer therapy adherence.

The information-motivation-behavioral skills (IMB) model, first proposed by Fisher, is composed of three elements-information, motivation, and behavioral skills-and is aimed at transferring patients' behavior into a positive direction, including self-behavior management ability, medication compliance and so on. For diabetic patients with poor adherence, the IMB model of care can be considered.

This model may be particularly useful in diabetic IOD patients since they are more prone to peri-implantitis than patients with other types of implant restorations or non-diabetic patients. However, the efficacy of the combination of the IMB model and continuity of care in improving healing, bone resorption, disease management and control, and quality of life in the specific population group of diabetic IOD patients remains unclear. To this end, the current study was aimed at investigating whether this model of care can help achieve better clinical outcomes and improve patient satisfaction with the services provided, thereby obtaining data to serve as a reference and scientific basis for the improvement of intervention plans.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria in this study were as follows:

1. IOD patients who had type 2 diabetes with peri-implantitis in at least one implant,
2. patients with clear consciousness and good communicative competence,
3. patients who could take good care of themselves and were proficient in using mobile communication and internet devices
4. patients who agreed to participate in our study.

Exclusion Criteria:

Patients with any of the following were excluded from our study:

1. type 1 diabetes and other particular types of diabetes,
2. severe cognitive dysfunction or psychiatric disorders, and
3. inability to use mobile electronic devices.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Peri-implant bone resorption | 1-2years
  Each patient received at least 3 panoramic radiographs on the first day patients came to our hospital for treatment of peri-implantitis (T0), 6 months after treatment (T1), and 12 months after treatment (T2), respectively. The distances from the most coronal implant-bone junction site to the implant platform in both the mesial and distal sites of the implants were measured and recorded as measured mesial bone level (mMBL) and measured distal bone level (mDBL) respectively. The lengths of the implants were measured in order to calibrate the measurements by using the actual known length of the implant, for example, the actual MBL(aMBL) = mMBL × (actual implant length) / (measured implant length). We obtained the average value of aMBL and aDBL, regarded T0 as the baseline, and subtracted T0 from T1 or T2 to acquire the bone loss in 6 or 12 months after treatment.

SECONDARY OUTCOMES:
Patient satisfaction | 1-2years
  An in-house questionnaire was developed to assess the patients' satisfaction regarding nurses service attitude, timeliness of responses, effectiveness in controlling peri-implant inflammation, and feelings about their own condition. The scores ranged from 1 to 10, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- The Stomatologic Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No